CLINICAL TRIAL: NCT05900232
Title: Anti KU Antibodies and Its Relationship With Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nehal Abdelbasset Ahmed, Resident Doctor at Rheumatology Department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-23-05-05MD
Record Dates: First submitted 2023-05-27; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anti _KU antibodies — aim of the work is to determine the relationship between Anti_Ku antibodies and SLE manifestations the study will include 60 SLE cases diagnosed by SLICC criteria and the activity of SLE will be calculated by SELDAI criteria, which is tool composed of 24 clinical and laboratory variables.

SUMMARY:
systemic lupus Erythematosus (SLE) is a multi system autoimmune disorder abroad spectrum of clinical presentations.

Diagnosis of SLE depending on Systemic Lupus International Collaborating Clinics (SLICC) Criteria.

SLICC Criteria requires either that a patient satisfy at least 4 of 17 Criteria including at least 1 of 11 clinical criteria and 1 of 6 immunological criteria or the patient has biopsy -proven nephritis compatible with SLE in the presence of antinuclear antibodies (ANA)or anti_double stranded DNA (dsDNA) antibodies.

Anti_KU antibodies included in (ANA), reported in many autoimmune disorders like SLE,Sjogren syndrome, idiopathic lung fibrosis and myositis.

So the aim of the work is to determine the relationship between Anti_KU antibodies and SLE manifestations.

ELIGIBILITY:
Inclusion Criteria:

* all patients will fulfill the Systemic Lupus International Clinics(SLICC) classification criteria for Systemic Lupus Erythematosus.

Exclusion Criteria:

* any patient with any collagen disease other than SLE

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Anti KU antibodies and its relationship with Systemic Lupus Erythematosus manifestations | 6 months
  the study will evaluate the titre of Anti KU
  antibodies which is positive or negative in one patient and on the other side what is the manifestation of SLE that found in the same patient if the Anti KU Antibodies titre is positive

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Egypt

REFERENCES:
- [Background] Mosca M, Bombardieri S. Assessing remission in systemic lupus erythematosus. Clin Exp Rheumatol. 2006 Nov-Dec;24(6 Suppl 43):S-99-104. PMID 17083771
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Background] Tsokos GC. Systemic lupus erythematosus. N Engl J Med. 2011 Dec 1;365(22):2110-21. doi: 10.1056/NEJMra1100359. No abstract available. PMID 22129255
- [Background] Mimori T. Clinical significance of anti-Ku autoantibodies--a serologic marker of overlap syndrome? Intern Med. 2002 Dec;41(12):1096-8. doi: 10.2169/internalmedicine.41.1096. No abstract available. PMID 12521194